CLINICAL TRIAL: NCT06943053
Title: Does Ioband Coverage Waterproof Dressing Provide Better Outcome Than Isolate Waterproof Dressing After Primary Total Knee Arthroplasty? A Prospective Randomized Controlled Trial
Brief Title: Evaluation of Ioband Coverage Waterproof Dressing Versus Isolated Waterproof Dressing After Primary Total Knee Arthroplasty
Acronym: Wound coverage
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Thammasat University Hospital (Other)
Responsible Party: Principal Investigator, Yot Tanariyakul, Krit Boontanapibul, Thammasat University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TUH wound coverage after TKA
Record Dates: First submitted 2025-04-09; First posted 2025-04-24 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Postoperative Wound Care After TKA
Keywords: total knee arthroplasty; Ioband® coverage waterproof dressing

STUDY DESIGN:
Intervention Model Description: Title: Evaluation of Ioband Coverage Waterproof Dressing Versus Isolated Waterproof Dressing After Primary Total Knee Arthroplasty
  Objective:
  -To compare the effectiveness of Ioband coverage waterproof dressing against traditional isolated waterproof dressing in terms of dressing performance, patient satisfaction, and wound management after primary total knee arthroplasty.
  Participants:
  * Total of 96 patients undergoing primary TKA.
  * Randomly assigned to two groups of 48 patients each:
  * Intervention Group: Ioband coverage waterproof dressing.
  * Control Group: Isolated waterproof dressing (Opsite®).
  Randomization Method:
  - Computerized block randomization conducted by an independent research assistant to ensure unbiased group allocation.
  Pre-operative protocol, surgical technique, post-operative pain control are the same
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control Group: Isolated waterproof dressing (Opsite®). (Active Comparator): Isolated waterproof dressing (Opsite®).
  Interventions: Device: Isolate waterproof dressing (Opsite)
- Ioban Coverage group (Experimental): Participants in this group will receive an Ioban iodine-impregnated antimicrobial incise drape placed over the standard water proof dressing at the end of primary total knee arthroplasty.the ioban drape extends 2 cm beyond the edge of the primary dressing and remain in place until dressing remove
  Interventions: Device: Ioban coverage group

INTERVENTIONS:
Device: Isolate waterproof dressing (Opsite) — Application of standard Opsite® waterproof dressing directly over the surgical incision following primary total knee arthroplasty. No additional drape or coverage was applied. The dressing remained in place until removal.
  Arms: Control Group: Isolated waterproof dressing (Opsite®).
Device: Ioban coverage group — Application of Ioban® iodine-impregnated antimicrobial incise drape over the standard waterproof dressing following primary total knee arthroplasty. The Ioban drape extends 2 cm beyond all edges of the dressing and remains in place until removal.
  Arms: Ioban Coverage group

SUMMARY:
Title: Evaluation of Ioband® Coverage Waterproof Dressing in Post-Operative Total Knee Arthroplasty (TKA)

Goal: To evaluate the effectiveness of Ioband® coverage waterproof dressing compared to standard waterproof dressing in reducing dressing change frequency and peel-off degree post-op TKA.

Main Research Questions:

1. Does Ioband® coverage waterproof dressing significantly decrease the degree of peel-off compared to standard waterproof dressing?
2. Does Ioband® coverage reduce the number of wound dressing changes required post-operatively?
3. Does Ioband® coverage improve overall patient satisfaction compared to standard waterproof dressing?

Participants:

Participants will include patients who have undergone total knee arthroplasty (TKA).

Main Tasks and Interventions:

1. Randomization: Participants will be randomly assigned to receive either the Ioband® coverage waterproof dressing or the standard waterproof dressing.
2. Application of Dressings: Participants will have the assigned dressing applied to their surgical site post-operatively.
3. Assessment of Peel-Off Degree: Participants will undergo assessments to evaluate the degree of peel-off of the dressing over a specified time.
4. Wound Dressing Changes: Participants will have their dressing changed as per routine care protocols, with documentation of the number of changes.
5. Patient Satisfaction Survey: Participants will complete a satisfaction survey to assess their experiences with the dressing and overall comfort.

Conclusion: The trial aims to provide insights into the benefits of Ioband® coverage waterproof dressing in improving post-operative care for TKA patients, focusing on key outcomes related to dressing performance and patient satisfaction.

DETAILED DESCRIPTION:
Study Design:

* Participants: 96 patients undergoing TKA, randomly assigned to two groups of 48 each:
* Intervention Group: Ioband® coverage waterproof dressing
* Control Group: Standard waterproof dressing (Opsite®)

Randomization Method:

-Computerized block randomization performed by an independent research assistant.

Pre-operative Procedures:

* Pre-emptive Analgesia administered 1 hour before surgery included:

  1. Naproxen (250 mg)
  2. Omeprazole (20 mg)
  3. Acetaminophen (500 mg)
  4. Pregabalin (75 mg)

     Anesthesia: Administered spinal anesthesia and ultrasound-guided adductor canal block by experienced anesthesiologists.

     Surgical Preparation:
* Incision sites were prepped and draped using sterile technique.
* Antiseptic Ioband® (60×45 cm) covered the incision site to prevent contamination.

Surgical Technique:

* Utilization of a standard medial parapatellar approach with a minimally invasive TKA technique.
* A tourniquet was inflated to 100 mmHg above systolic blood pressure and was deflated after wound closure.
* Cemented posterior stabilizer prosthetics (Nexgen LPS) and patellar resurfacing were used.
* Anesthetic cocktail (0.5% bupivacaine, adrenaline, ketorolac, morphine) was injected around the capsule after prosthesis insertion.

Post-operative Care:

* No suction drains or extremity wraps used.
* Wounds closed with waterproof dressing (Opsite® size 25×10 cm) in 90-degree knee flexion without tension.
* Pain Management: Multimodal pain control was employed.
* Antibiotic Prophylaxis: Administered for 24 hours post-surgery.
* Rehabilitation: Early knee range of motion exercises and ambulation were encouraged within 24 hours post-operation.

Wound Management Protocol:

* Patients were allowed to start bathing 48 hours post-op.
* Dressing change on post-op day 3, using sterile technique:
* Control Group: Covered with waterproof dressing (Opsite®).
* Intervention Group: Covered with Ioband® in knee flexion.

Wound Care Instructions:

* Keep covering material dry and clean; avoid irritation.
* Report any signs of infection (redness, swelling, fever) to a doctor.
* Avoid creams or powders unless prescribed.
* Avoid scratching or rubbing around the wound.
* Light activities permitted; avoid strenuous activities for 6 weeks.
* Dressing should not be changed until advised, typically after 14 days unless signs of complications are observed.

Criteria for Dressing Change:

* Change dressing if:
* First waterproof dressing peels off grade II or III.
* Second dressing has over 50% bleeding.
* Suspected surgical site infection. Patients were also included in a chat group for wound care consultation.

ELIGIBILITY:
Inclusion Criteria:

* Primary unilateral TKA
* Age 55-80 yrs

Exclusion Criteria:

* Chronic Skin disease such as Psoriasis
* Chronic steroid use
* Allergy to skin adhesive, Cover wound
* Robotic TKA
* Iodine allergy
* Not follow protocol

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2025-04-06 (Actual); Primary Completion 2026-04-06 (Estimated); Study Completion 2026-04-16 (Estimated)

PRIMARY OUTCOMES:
Number of change wound dressing | 14 days postoperation
  Indication for changing wound dressing before appointment
  1. Post op wound with waterproof peel off grade II (waterproof peel off to pad) or grade III (waterproof peel off involve into pad)
  2. Waterproof has bloody more than 50 %
  3. suspected Surgical site infection

SECONDARY OUTCOMES:
Degree of peel off wound | 14 days postoperation
  There are 4 types of Characteristics of the Wound Sealant Leakage Level 0: No leakage of the plastic sealant. No need to open the wound Level 1: Plastic sealant leaks around the edges but not into the wound. No need to open the wound Level 2: Plastic sealant leaks around the edges up to the wound edge. Open the wound and re-seal with a new sealant Level 3: Plastic sealant leaks deep into the wound edges. Open the wound and re-seal with a new sealant
Satisfactory of patient | 14 days post-operation
  * Satisfactory of patient: (score1-10)
  * Comfort for wound care (score 0-10)
  * Difficult to take a bath (score 0-10)
  * Pain on remove dressing (score 0-10)
  * Cost for Dressing after D/C
Post op Range of motion of knee | At 2 weeks, 6 weeks and 3 months postoperation
  Degree of flexion
Wound-related Complication | At 2 weeks, 6 weeks and 3 months postoperation
  Wound-related Complication
  * Skin bleb, redness
  * Dehiscence
  * Subcutaneous hematoma
  * Surgical site infection

CONTACTS AND LOCATIONS:
Overall Officials: Chanon Thassanaleelaporn, M.D., Principal Investigator — Thammasat University Hospital Thailand; Krit Boontanapibul, M.D., Study Director — Thammasat University Hospital
Locations (2):
- Thailand (2):
  - Thammasat University Hospital, Pathum Thani, Khlong luang
  - Department of Orthopaedics, Thammasat University, Pathum Thani

IPD SHARING:
Plan to Share IPD: No
The datasets analyzed during the current study are not available due to protect study participant privacy.

REFERENCES:
- [Background] 1 Primary Total Knee Replacement: A Recipe for Dry Dressing Azfar KM, Adil AO, Tarig AR, Adel G. Primary Total Knee Replacement: A Recipe for Dry Dressing. Cureus. 2023;15(4). 2 The effect of different wound dressing materials used in postoperative treatment of wounds after total hip arthroplasty and total knee arthroplasty: A meta-analysis Yingjia Yuan, Jin Li, Ke Wang, Guanqiang Zheng, Shengting Chai. The effect of different wound dressing materials used in postoperative treatment of wounds after total hip arthroplasty and total knee arthroplasty: A meta-analysis.IWJ. : April 2022. 3 Clinical outcome of different skin closure in TKA Chen L, Yang J, Xie J, Hu Y, Zeng M. Clinical outcome of different skin closure in total-knee arthroplasty: running subcuticular closure vs intermittent closure: a retrospective study. Medicine. 2020 Aug 8;99(34). 4 Closure in knee replacement surgery Kharat K. Closure in knee replacement surgery. Journal of Orthopaedic Case Reports. 2012 Jul;2(3):31. 5 Multilayer watertight closure to address adverse event from primary total knee and hip arthroplasty Snyder MA, Chen BP, Hogan A, Wright GW. Multilayer watertight closure to address adverse events from primary total knee and hip arthroplasty: a systematic review of wound closure methods by tissue layer. Arthroplasty today. 2021 Aug 1;10:180-9. 6 Persistent wound drainage after total joint arthroplasty: a narrative review Wagenaar FC, Löwik CA, Zahar A, Jutte PC, Gehrke T, Parvizi J. Persistent wound drainage after total joint arthroplasty: a narrative review. The Journal of Arthroplasty. 2019 Jan 1;34(1):175-82. 7 Effect of the knee position during wound closure after TKA on early knee function recovery. Wang S, Xia J, Wei Y, Wu J, Huang G. Effect of the knee position during wound closure after total knee arthroplasty on early knee function recovery. Journal of Orthopaedic Surgery and Research. 2014 Dec;9(1):1-6